CLINICAL TRIAL: NCT02182960
Title: An Open Two Way Cross Over Study to Relative Bioavailability of Ibuprofen Enantiomers After Single p.o. Administration of 200 mg Syrup (T) Compared With 200 mg Standard Brufen Sirup (R)
Brief Title: Bioavailability of Ibuprofen Enantiomers Compared With Standard Brufen Sirup in Healthy Male Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 1024.3
Record Dates: First submitted 2014-07-04; First posted 2014-07-08 (Estimated); Last update posted 2018-08-31 (Actual); Status verified 2018-08

CONDITIONS: Healthy

ARMS (2):
- Ibuprofen (Experimental)
  Interventions: Drug: Ibuprofen syrup
- Brufen (Active Comparator)
  Interventions: Drug: Brufen syrup

INTERVENTIONS:
Drug: Ibuprofen syrup
  Arms: Ibuprofen
Drug: Brufen syrup
  Arms: Brufen

SUMMARY:
Pharmacokinetics (relative bioavailability), safety and tolerability

ELIGIBILITY:
Inclusion Criteria:

* Healthy males from 21 to 50 years and within +-20% of their normal weight (Broca index)
* Written informed consent

Exclusion Criteria:

* Any findings of the medical examination or laboratory tests deviating from normal and of clinical relevance
* Gastrointestinal, hepatic, renal, respiratory (especially bronchial asthma and chronic obstructive pulmonary disease), cardiovascular, metabolic, immunological or hormonal disorders
* Diseases of the central nervous system (such as epilepsy) or psychiatric disorders
* History of orthostatic hypotension, fainting spells or blackouts
* Chronic or relevant acute infections
* History of allergy/hypersensitivity (including drug allergy) which is deemed relevant to the trial as judged by the investigator
* Intake of a drug with a long half-life (>=24 hours) within at least one month or less than ten half-lives of the respective drug before enrolment in the study
* Use of any drugs which might influence the results of the trial within seven days prior to administration or during the trial
* Participation in another trial with an investigational drug within two months prior to the start of the study
* Smoker (> 10 cigarettes or 3 cigars or 3 pipes/day)
* Inability to refrain from smoking on study days
* Alcohol abuse
* Drug abuse
* Blood donation (>100 ml) within four weeks prior to administration
* Other disease or abnormality of clinical relevance
* Excessive physical activities within two weeks prior to administration or during the trial

Ages: 21 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 1998-09; Primary Completion 1998-10 (Actual)

PRIMARY OUTCOMES:
Total area under the plasma drug concentration-time curve from time zero to infinity (AUC0-∞) | Up to 12 hours after each administration
Maximum drug plasma concentration (Cmax) | Up to 12 hours after each administration

SECONDARY OUTCOMES:
Time to reach the maximum concentration of the analyte in plasma (tmax) | Up to 12 hours after each administration
Apparent terminal rate constant (λz) | Up to 12 hours after each administration
Apparent terminal half-life of the analyte in plasma (t1/2) | Up to 12 hours after each administration
Total area under the plasma drug concentration-time curve from time zero to the last quantifiable drug (AUC0-t(last)) | Up to 12 hours after each administration
Mean residence time, total (MRTtot) | Up to 12 hours after each administration
Total plasma clearance divided by the systemic availability factor (CL/f) | Up to 12 hours after each administration
Volume of distribution during the terminal phase λz, divided by f (Vz/f) | Up to 12 hours after each administration
Number of adverse events | Up to 8 days after last drug administration
Change from baseline in 12-lead ECG (electrocardiogram) | Baseline, 8 days after last drug administration
Change in vital functions (blood pressure and puls rate) | Baseline, up to 8 days after last drug administration
Change from baseline in standard laboratory evaluation | Baseline, 8 days after last drug administration